CLINICAL TRIAL: NCT05223270
Title: The Effect of Different Wound Dressing on Prevention of Pressure Injury Related to Noninvasive Mechanical Ventilation Mask in Patients With Respiratory Failure
Brief Title: the Effect of Different Wound Dressing on Prevention of Pressure ınjury Related to NIMV Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, pınar dogan, Asst.Prof., Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1019181716
Record Dates: First submitted 2021-08-16; First posted 2022-02-03 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Pressure Injury
Keywords: noninvasive mechanical ventilation; pressure injury; wound dressing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: semi-experimental study with post test, control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group-1 (Experimental): Hydrocolloid wound dressings were placed on the pressure areas under the NIMV mask of the patients in this group.
  Interventions: Other: wound dressing under the NIMV mask
- intervention group-2 (Experimental): Hydrocelluler wound dressings were placed on the pressure areas under the NIMV mask of the patients in this group.
  Interventions: Other: wound dressing under the NIMV mask
- control group (No Intervention): Patients in this group were treated without placing an additional dressing under the NIMV mask.

INTERVENTIONS:
Other: wound dressing under the NIMV mask — wound dressing under the NIMV mask
  Arms: intervention group-1; intervention group-2

SUMMARY:
This study is aimed to examine the effect of different wound dressings on the prevention of pressure injury in the face area related to noninvasive mechanical ventilation mask. The study was completed out with 102 patients who were followed up in Chest Diseases and Thoracic Surgery Hospital between October 2019 and August 2020 and met the inclusion criteria of the study. In the study, hydrocellular and hydrocolloid wound dressing was applied to the pressure areas under the mask of noninvasive mechanical ventilation in the intervention groups, while the routine treatment process was followed in the control group. Wound dressings were obtained from HARTMANN. Study data were collected with the "Individual Characteristics Form" and "Pressure Injury Rating Scale".

DETAILED DESCRIPTION:
In the hospital where the study was conducted, patients with respiratory failure receive NIMV treatment with an oro-nasal mask. In the study, hydrocolloid and hydrocellular wound dressings were placed on the pressure areas under the mask of the patients in the intervention group. NIMV treatment was applied to the face area of the patients in the control group with an oronasal mask without using any barrier cover. The pressure areas of the patients in the intervention and control groups were evaluated with the pressure injury scale before and after the NIMV treatment. Follow-up was carried out twice a day for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years, receiving NIMV therapy for at least 6 hours a day, on the first day of hospitalization and followed up for at least 7 days, receiving NIMV treatment with an oro-nasal mask, tolerant of mask,

Exclusion Criteria:

* patients with pre-treatment pressure injuries in the facial area, patients with diabetes mellitus, patients with mental or psychological problems

Ages: 22 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
pressure injury stage | 1st day
  The development of pressure injury in the facial region of the patients after the intervention was evaluated twice a day with the pressure injury scale.
pressure injury stage | 2nd day
  The development of pressure injury in the facial region of the patients after the intervention was evaluated twice a day with the pressure injury scale.
pressure injury stage | 3rd day
  The development of pressure injury in the facial region of the patients after the intervention was evaluated twice a day with the pressure injury scale.
pressure injury stage | 4th day
  The development of pressure injury in the facial region of the patients after the intervention was evaluated twice a day with the pressure injury scale.
pressure injury stage | 5th day
  The development of pressure injury in the facial region of the patients after the intervention was evaluated twice a day with the pressure injury scale.
pressure injury stage | 6th day
  The development of pressure injury in the facial region of the patients after the intervention was evaluated twice a day with the pressure injury scale.
pressure injury stage | 7th day
  The development of pressure injury in the facial region of the patients after the intervention was evaluated twice a day with the pressure injury scale.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Dogan, Asst.Prof., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It will be presented as a Clinical Study Report.
Supporting Information: CSR
Time Frame: It will be used in the period from the completion of the study to the publication of the article (average 15 months).
Access Criteria: Supporting meta-analysis studies that need the data of the study can be shared.